CLINICAL TRIAL: NCT05513144
Title: Monitoring Circulating Tumor DNA and Evaluating Prognostic and Predictive Impact of Liquid Biopsy in Advanced HER2 Negative Gastric Cancer
Brief Title: Potential Clinical Utilities of Circulating Tumor DNA in Advanced HER2 Negative Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: chenwu (Other)
Responsible Party: Sponsor-Investigator, chenwu, Department of Oncology, The First People's Hospital of Changzhou
Organization: The First People's Hospital of Changzhou (Other)
Other Study IDs: 2022-CL048-01
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer; Circulating Tumor DNA (ctDNA)
Keywords: Gastric Cancer; Circulating Tumor DNA; Prognosis; Therapy Response
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the use of next generation sequencing (NGS) to detect circulating tumor DNA in advanced HER2 negative gastric cancer patients. The evaluation of the therapy efficacy for gastric cancer patients is usually evaluated by computer tomography scans with RECIST criteria that are performed every two months during the treatment. In this study, we will compare the monitoring of circulating tumor DNA with the results of CT scan according the RECIST criteria and the blood level of CEA and CA 19-9 tumor markers.

DETAILED DESCRIPTION:
Gastric cancer is one of the common malignant tumors in China, with relatively high incident rate and mortality among the population. More than 80% of gastric cancer are in advanced stage.

Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 166 bp, mixed with cell free DNA (cfDNA) of other sources in blood circulation.ctDNA is reflecting the most up-to-date status of tumor genome. Hence, it is considered as a new biomarker for tumor, which can be qualitative, quantitative and used for disease monitoring. Detecting ctDNA, in most patients, allows for the noninvasive molecular characterization detection of tumors, including genetic changes that are revealed by the selective pressure of therapies. Considering the origin of ctDNA, it can be from different subclones of primary tumor or both primary and metastatic tumors, the ctDNA may overcome the problems caused by tumor heterogeneity. Additionally, the short half-life of ctDNA, about 2 hours, makes ctDNA an ideal dynamic marker of tumor bulk.

Molecular events including gene mutation, fusion and amplification will be detected by next generation sequencing platform using ctDNA collected from peripheral blood samples of gastric cancer patients. Samples will be collected at baseline, every two months in the surveillance after treatment and disease progression.

Thus, the objective of this study is to identify a prognostic and/or predictive biomarker of tumor response according to the tumor DNA circulating assessment in gastric cancer treatment, in order (i) to avoid an unnecessary toxicity of an ineffective treatment that it would be continued uselessly, (ii) and to allow a early changing to an alternative therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 - 75.
2. Histologically confirmed adenocarcinoma of gastric or gastro-oesophageal junction. Gastric tumors should be treatment naïve unresectable or metastatic disease, or recurrence over 6 months after finish of adjuvant chemotherapy.
3. HER2 status is confirmed by IHC/FISH. HER2 negative: IHC 0/1+ or IHC 2+ plus FISH negative.
4. At least one measurable lesion should be confirmed by imaging examination.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. No concomitant other malignant tumor or treated malignant tumor within last five years.
7. Eligible peripheral blood and tissue samples.
8. Willing to provide clinicopathological information and imaging information.

Exclusion Criteria:

1. Patients received systemic treatment before enrolled or finished adjuvant chemotherapy less than 6 months.
2. With second primary malignant diseases.
3. HER2 status is confirmed by IHC/FISH. HER2 positive: IHC 3+ or IHC 2+ plus FISH positive.
4. No qualified paired tissue samples.
5. No complete clinicopathological information and follow-up.
6. Presence of any systemic illness incompatible with participation in the clinical trial or inability to provide written informed consent.
7. Other situations assessed by investigator can disturb quality control of the investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 negative gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Prognostic molecular markers. | 2 years
  Change from baseline in molecular biomarkers at time on disease progression
The sensitivity and specificity of ctDNA detection. Profiling of the most frequently detected gene mutations and level of mutations in ctDNA | 2 years

SECONDARY OUTCOMES:
Mutation profile and the concordance of mutations in tumor tissue and ctDNA of gastric cancer | 2 years
Mechanisms of therapy resistance | 2 years
  Screening out the molecular markers related to the therapy resistance of gastric cancer by comparing molecular profiles on baseline and disease progression of patients with different therapy response
The concordance and accuracy of response evaluation results determined by ctDNA compared with imaging and serum tumor biomarkers (CEA, CA19-9,CA72-4 et al). | 2 years
Relative frequency of targetable mutations (incl. TMB and MSI status). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China